CLINICAL TRIAL: NCT05914792
Title: Longitudinal ctDNA Monitoring in Older Women With ER+ Breast Cancer Who Forego Upfront Surgery in Favor of Primary Endocrine Therapy
Brief Title: Longitudinal ctDNA Surveillance for Older Women With ER+ Breast Cancer Who Omit Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Principal Investigator, Priscilla McAuliffe, Assistant Professor of Medicine, University of Pittsburgh
Other Study IDs: HCC 22-088; STUDY21100091 (Other: University of Pittsburgh)
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: estrogen receptor positive (ER+); progesterone receptor (PR+); early-stage breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient blood to track ctDNA longitudinally over time as well as any tissue samples that the patient may have (including core biopsy samples and/or surgical specimens should the patient and their treating physician decide to undergo salvage surgery at any point).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective study recruits patients with ER+/HER2-, non-metastatic breast cancer who omit upfront surgery in favor of primary endocrine therapy for sample collection and prospective circulating tumor DNA (ctDNA) measurement to guide disease surveillance.

DETAILED DESCRIPTION:
Age is one of the most important risk factors for the development of breast cancer. Nearly a third of all breast cancer cases occur in older women (aged ≥ 70 years), with most cases being estrogen receptor-positive (ER+). Such tumours are unlikely to be the ultimate cause of death for older women, particularly when considering other comorbidities. Our group has recently shown that risk of breast cancer-related mortality is only around 3% for older women who forego upfront surgery and instead treated with primary endocrine monotherapy. However, with omission of surgery, surveillance for tumor growth or treatment failure is important but requires patients (and their caregivers) to have regular imaging and to see their oncology team every 3 months, which can be quite burdensome. Thus, this study employs a ctDNA surveillance scheme to monitor for potential tumor growth. Partnering with Natera, this study uses a bespoke, tumor-specific ctDNA assay (Signatera) to monitor for changes in ctDNA dynamics while the patient is on endocrine therapy.

This study is for patients who choose not to undergo primary surgical intervention and are managed medically on primary endocrine therapy (any endocrine therapy permitted). Patients will undergo Signatera testing at the time of regularly scheduled clinic follow-up visits and/or at the time of surveillance imaging, which will occur every 3-6 months. Patients will also be asked to complete regular surveys while participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* early-stage (stages I-III) breast cancer
* estrogen receptor positive (ER+) and/or progesterone receptor positive (PR+) and HER2 receptor negative
* able to provide blood samples
* decision made by treating physician and patient to forego upfront surgery in favor of medical management with endocrine therapy
* non-metastatic disease at diagnosis (patients need not have staging scans; patients at higher risk for de novo stage IV disease should not have any symptoms concerning for metastatic disease)
* patients may be taking any endocrine therapy
* patients may be taking any CDK4/6 inhibitor as deemed necessary by their treating physician
* any ECOG Performance Status allowed
* if patients have synchronous bilateral ER+ breast cancer, tissue from both sites should be submitted to Natera to perform ctDNA testing
* patients with multifocal/multicentric tumors are eligible and the largest focus of cancer should be submitted for testing

Exclusion Criteria:

* under 70 years of age
* breast cancer that is not estrogen receptor positive (ER+) or progesterone receptor (PR+)
* unable to provide blood samples or insufficient tumor tissue for Signatera testing

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Women only with ER+ breast cancer
Study Population: Women 70 years of age or older with ER+/HER2-, non-metastatic breast cancer who forego upfront surgery in favor of primary endocrine therapy.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of ctDNA positivity | Up to 5 years
  Proportion of patients with ER+/HER2- breast cancer who omit upfront surgery in favor of primary endocrine therapy who have any ctDNA positivity using Signatera assay.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years
  The length of time after treatment initiation that patient is alive and without any evidence of tumor progression as defined by RECIST1.1 criteria. Per RECISIT v1.1: Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Breast cancer-specific survival (BCSS) | Up to 5 years
  BCSS is defined as the length of time from the date of diagnosis through the end of follow up that patients are free from breast cancer-related mortality.
Overall survival (OS) | Up to 5 years
  The length of time from the date of diagnosis through the end of follow up that patients are still alive.
Longitudinal quality of life assessment using National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Breast Cancer Symptom Index - 16 Item Version (NCCN NFBSI-16) | Up to 5 years
  This assessment is a 16 item questionnaire using Likert scale (0-4) measured with each ctDNA blood draw. Score ranges from 0-64 with higher scores indicative of higher quality of life / asymptomatic from cancer-related therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla McAuliffe, MD, PhD, Principal Investigator — UPMC Magee Women's Hospital, UPMC Hillman Cancer Center
Locations (1):
- UPMC Magee Womens Hospital - Surgical Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No